CLINICAL TRIAL: NCT03918993
Title: Evaluation of the Effects of a Daily Dose of 5 mg of Tadalafil on Lymphocyte to Monocyte Ratio and Monocyte to High-Density Lipoprotein Ratio in Patients With Erectile Dysfunction
Brief Title: Effects of Tadalafil on LMR and MHR in Patients With ED
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Mehmet Necmettin Mercimek, Principal Investigator, Samsun Liv Hospital
Other Study IDs: OMU KAEK 2019/158
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Erectile Dysfunction; Inflammation
Keywords: Erectile Dysfunction; lymphocyte to monocyte ratio; monocyte to HDL ratio
MeSH Terms: conditions — Erectile Dysfunction; Inflammation | interventions — Tadalafil; Tablets; Cyclic Nucleotide Phosphodiesterases, Type 5; PDE5A protein, human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group T: 31 Patients with ED who receiving 5 mg/day of Tadalafil for 8 weeks.
  Interventions: Drug: Tadalafil 5mg tablet
- Group C: Thirty-one healthy men who were admitted to the internal medicine outpatient clinic for their annual follow-up

INTERVENTIONS:
Drug: Tadalafil 5mg tablet — Once-a-day 5 mg dose of tadalafil for 8 weeks
  Other Names: phosphodiesterase type 5 (PDE5) inhibitor
  Groups: Group T

SUMMARY:
The aim of the study was to investigate whether daily 5 mg tadalafil over eight weeks affects to Lymphocyte/Monocyte ratio (LMR) and Monocyte/High-Density Lipoprotein ratio (MHR) in patients with erectile dysfunction (ED).

Thirty-one patients with organic ED and 31 healthy controls between July 2017 and November 2018 were included in this retrospective study. To avoid bias, the patients were randomly selected and the controls were also incorporated consecutively. The presence of ED was determined according to the International Erectile Function Index-5 (IIEF-5). The patients and the controls were evaluated in terms of IIEF-5, complete blood count, serum biochemistry, LMR, and MHR.

DETAILED DESCRIPTION:
The medical records of the heterosexual men treated with the diagnosis of organic ED in the Urology department of a private hospital between July 2017 and October 2018 were evaluated retrospectively. The number of samples to be included in the study was determined by the help of the computer-assisted power analysis. Random sampling was performed from all cohorts of patients with ED. Thirty-one male patients between the ages of 39-65 with organic erectile dysfunction more than one year and treated with OAD 5 mg dose of tadalafil for eight weeks were selected as the treatment group (group T)The patients in group T have been assessed both before (T1) and after (T2) the treatment.

Between the ages of 39-65, thirty-one healthy men who were admitted to the internal medicine outpatient clinic for their annual follow-up were selected consecutively and the control group (group C) was formed. All subjects in the control group were sexually active men with regular monogamous heterosexual relationships during the last one year.

.

ELIGIBILITY:
Inclusion Criteria:

* 39-65 years old men with ED
* 39-65 years old, haelthy men
* Patients that have received 5 mg tadalafil/day for 8 weeks
* Patients with informed consent forms
* Patients with no missing variables

Exclusion Criteria:

* Patients with systemic autoimmune and inflammatory disease,
* congestive heart failure,
* chronic renal failure, and chronic hepatobiliary disease,
* chronic lung disease, and thyroid dysfunction,
* patients with acute infection,
* patients with neurological deficits,
* metabolic syndrome and malignancy
* Patients with a history of prostate, penile or pelvic surgery or radiotherapy,,
* patients receiving anticoagulant, beta-blocker, antidepressants and antipsychotics, hormonal therapy,
* patients with alcohol and smoking

Ages: 39 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between the ages of 39-65, thirty-one healthy men who were admitted to the internal medicine outpatient clinic for their annual follow-up were selected consecutively and the control group Thirty-one male patients with organic erectile dysfunction more than one year between 39 and 65 years of age which were treated with OAD 5 mg dose of tadalafil for eight weeks were selected as the treatment group
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Lymphocyte to Monocyte Ratio | up to 8 weeks
  ratio of values in complete blood count
monocyte to HDL ratio | up to 8 weeks
  an inflamamtoy marker
The International Index of Erectile Function (IIEF-5) Questionnaire | up to 8 weeks
  IIEF-5 scoring:
  The IIEF-5 score is the sum of the ordinal responses to the 5 items. 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunctio
monocyte count | up to 8 weeks
  complete blood count
lymphocyte count | up to 8 weeks
  complete blood count
HDL cholesterol | up to 8 weeks
  serum lipid profile
Testosteron | up to 8 weeks
  hormonal evaluation
fasting glucose | at the 1st day
  serum glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Yakup Bostancı, MD, Study Chair — Ondokuz Mayıs University
Locations (1):
- Samsun Liv Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta BP, Murad MH, Clifton MM, Prokop L, Nehra A, Kopecky SL. The effect of lifestyle modification and cardiovascular risk factor reduction on erectile dysfunction: a systematic review and meta-analysis. Arch Intern Med. 2011 Nov 14;171(20):1797-803. doi: 10.1001/archinternmed.2011.440. Epub 2011 Sep 12. PMID 21911624
- [Result] Kadihasanoglu M, Karabay E, Yucetas U, Erkan E, Ozbek E. Relation between Monocyte to High-Density Lipoprotein Cholesterol Ratio and Presence and Severity of Erectile Dysfunction. Aktuelle Urol. 2018 Jun;49(3):256-261. doi: 10.1055/s-0042-123163. Epub 2017 Nov 16. PMID 29145685
- [Result] Cimen S, Dursun M, Sulukaya M, Besiroglu H. Could the monocyte/HDL cholesterol ratio be an early marker of erectile dysfunction? Aging Male. 2020 Dec;23(5):694-699. doi: 10.1080/13685538.2019.1574735. Epub 2019 Feb 19. PMID 30777468